CLINICAL TRIAL: NCT06649422
Title: Clinical Study on the Efficacy and Safety of Reduced-Dose Chemotherapy Followed by 14 Days of Blinatumomab in Adult Patients with Newly Diagnosed Ph-Negative B-ALL: a Prospective, Multicenter, Observational Study.
Brief Title: Reduced-Dose Chemo Followed by 14 Days of Blinatumomab for Newly Diagnosed Adult B-ALL Patients: a Multicenter Study
Status: Not yet recruiting | Type: Observational
Sponsor: Shandong University (Other)
Collaborators: Shandong Provincial Hospital (Other Government); The Affiliated Hospital of Qingdao University (Other); Tangshan Central Hospital (Other); Affiliated Central Hospital of Shandong First Medical University (Unknown); Yantai Yuhuangding Hospital (Other); Qilu Hospital of Shandong University (Qingdao) (Other); Qingdao Central Hospital (Other); Qingdao Municipal Hospital (Other); The Affiliated Hospital of Jining Medical University and Zaozhuang City (Unknown); Affiliated Hospital of Binzhou Medical College (Unknown); Linyi People's Hospital (Other); The Second Hospital of Shandong University (Other); Affiliated Hospital of Shandong University of Traditional Chinese Medicine (Other); Shandong First Medical University (Other); Shengli Oilfield Hospital (Other); Heze Municipal Hospital (Other); Zibo Central Hospital (Other Government); Zaozhuang Municipal Hospital (Other); Weihai Municipal Hospital (Other)
Responsible Party: Principal Investigator, Chunyan Ji, Prof., Qilu Hospital of Shandong University
Other Study IDs: QLCR20240289
Record Dates: First submitted 2024-09-06; First posted 2024-10-18 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-07

CONDITIONS: Leukemia, Lymphocytic, Acute, Adult
Keywords: blinatumomab; newly diagnosed Ph-chromosome negative acute B-lymphoblastic leukemia; induction treatment; reduced-dose chemotherapy
MeSH Terms: conditions — Leukemia | interventions — blinatumomab; Drug Therapy, Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Reduced-dose chemotherapy followed by blinatumomab induction treatment group: Patients aged 15-65 with newly diagnosed Ph-negative B-ALL undergoing frontline induction therapy with reduced-dose chemotherapy followed by blinatumomab.
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — The 14-day blinatumomab combined with reduced-dose chemotherapy is used for the induction treatment of newly diagnosed Ph-chromosome negative acute B-lymphoblastic leukemia.
  Other Names: Combination chemotherapy with multiple drugs.; preventive intrathecal injections

SUMMARY:
This is a prospective, multicenter, observational study aimed at exploring the efficacy and safety of reduced-dose chemotherapy followed by frontline therapy with blinatumomab in patients aged 15-65 with newly diagnosed Ph-negative B-ALL.

DETAILED DESCRIPTION:
The 14-day blinatumomab combined with reduced-dose chemotherapy is used for the induction treatment of newly diagnosed Ph-chromosome negative acute B-lymphoblastic leukemia. On day 14, an intrathecal injection of chemotherapy is administered; on days 28-35, bone marrow is assessed, and patients who do not achieve complete remission are withdrawn from the study. Patients with positive minimal residual disease (MRD) after induction treatment undergo transplant typing and proceed to allogeneic hematopoietic stem cell transplantation (Allo-HSCT) after early intensification. Patients with negative MRD receive alternating treatment with multi-drug combination chemotherapy and blinatumomab, for a total of 8 consolidation courses, including 3 courses of blinatumomab. Maintenance therapy lasts for at least 18 months, using the POMP regimen with or without one cycle of blinatumomab every six months. Throughout the entire treatment phase, at least 12 preventive intrathecal injections are administered.

ELIGIBILITY:
Inclusion Criteria:

* Age 15-65 years, both male and female are eligible;
* Untreated newly diagnosed Ph-negative B-ALL patients; Diagnosis is defined by using morphological, immunological, cytogenetic, and molecular (MICM) diagnostic models, with immunotyping showing >20% primitive lymphoid cells in the bone marrow; bone marrow cytogenetics showing Philadelphia chromosome (Ph) negative (after observing at least 20 metaphases) and/or fluorescence in situ hybridization (FISH) BCR/ABL negative and/or molecular BCR/ABL fusion gene negative;
* Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-2;
* Organ function tests must meet all the following criteria: Total bilirubin <1.5×upper limit of normal (ULN); Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST) <2.5×ULN (if liver is involved, then ALT and AST <5×ULN are allowed); Creatinine <1.5×ULN; Serum amylase and lipase ≤1.5×ULN; Alkaline phosphatase ≤2.5× ULN; Serum electrolytes potassium, magnesium, phosphorus within normal limits.
* Cardiac color Doppler echocardiography ejection fraction ≥45%;
* Female patients of childbearing potential must have a negative pregnancy test (within 7 days prior to enrollment).

Exclusion Criteria:

* Previous or ongoing systemic anti-acute lymphoblastic leukemia (ALL) treatment (including but not limited to radiotherapy), except for appropriate pretreatment;
* Clinical manifestations of central nervous system or extramedullary involvement at the time of diagnosis;
* Patients participating in other clinical studies simultaneously;
* Accompanying diseases that, in the judgment of the investigator, pose a serious risk to patient safety or affect the patient's ability to complete the study;
* A history of definite neurological or psychiatric disorders, including epilepsy or dementia;
* Major surgery within the last 4 weeks or not recovered from previous surgery;
* Having other malignant tumors, unless the other primary malignant tumor is currently stable or does not require active intervention;
* Women of childbearing age or men who cannot use sufficient methods for contraception, including pregnant or lactating women;
* Clinically significant severe uncontrollable heart disease (including but not limited to a history of myocardial infarction, stroke, or revascularization; unstable angina or transient ischemic attack within 6 months before enrollment; congestive heart failure or left ventricular ejection fraction (LVEF) below the local institutional standard lower limit within 6 months before enrollment; a history of clinically significant (determined by the attending physician) atrial arrhythmia; a history of ventricular arrhythmia; a history of venous thromboembolism, including deep vein thrombosis or pulmonary embolism, uncontrollable hypertension, etc.);
* Confirmed positive status for human immunodeficiency;
* Active severe infections that cannot be controlled by oral or intravenous antibiotics;
* Patients known to be allergic or contraindicated to the study drug (active pharmaceutical ingredient and/or excipients);
* Existence of bleeding disorders unrelated to ALL.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 15-65 years newly diagnosed with Philadelphia chromosome-negative acute B-lymphoblastic leukemia, confirmed at Qilu Hospital of Shandong University and other participating institutions in Shandong Province.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
The overall response rate | At the end of induction treatment from day 28 to day 35
  The overall response rate after induction therapy = Complete Remission (CR) + CR with partial hematologic recovery (CRh) + CR with incomplete hematologic recovery (Cri).
Minimal Residual Disease (MRD) negativity rate after induction therapy | At the end of induction treatment from day 28 to day 35
  MRD negativity refers to a flow cytometry test result where MRD is less than 0.01%.

SECONDARY OUTCOMES:
Complete molecular remission rate. | At the end of induction treatment from day 28 to day 35
  Complete molecular remission rate is defined as undetectable Ig rearrangement by next-generation sequencing, with a detection sensitivity of at least less than 10^-5.
One-year overall survival rate. | From diagnosis of the disease to the end of the first year
  The proportion of patients who are still alive one year after the date of disease diagnosis, out of the total number of subjects enrolled in the study.
One-year event-free survival rate | From diagnosis of the disease to the end of the first year
  The proportion of patients who have not experienced disease progression, been diagnosed with another cancer, or died from any cause one year after the date of disease diagnosis, out of the total number of subjects enrolled in the study.
Safety | From enrollment until withdrawal from the study or the end of follow-up up to two years
  Safety endpoints are defined, graded, and evaluated according to the CTCAE version 5.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Chunyan Ji, Doctor, Principal Investigator — Qilu Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: Undecided